CLINICAL TRIAL: NCT03295721
Title: A Phase 3, Randomized, Double Blind, Saline Placebo and Active Controlled, Multicenter Study of HTX 011 Via Local Administration for Postoperative Analgesia and Decreased Opioid Use Following Unilateral Simple Bunionectomy
Brief Title: Bunionectomy Study for Postoperative Analgesia (EPOCH 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HTX-011-301
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain
Keywords: bunion; bunionectomy; bunion surgery; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Bunion | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Treatment Group 1: HTX-011 (Experimental): HTX 011 (bupivacaine/meloxicam)
  Interventions: Drug: HTX-011; Device: Luer-lock applicator; Device: Vial access device
- Treatment Group 2: Saline Placebo (Placebo Comparator): Saline placebo
  Interventions: Drug: Saline Placebo; Device: Luer-lock applicator
- Treatment Group 3: Bupivacaine HCI (Active Comparator): Bupivacaine HCl
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: HTX-011 — HTX 011 (bupivacaine/meloxicam), 60 mg/1.8 mg by instillation
  Arms: Treatment Group 1: HTX-011
Drug: Saline Placebo — Saline placebo by instillation
  Arms: Treatment Group 2: Saline Placebo
Drug: Bupivacaine HCl — Bupivacaine HCl without epinephrine, 50 mg by injection
  Arms: Treatment Group 3: Bupivacaine HCI
Device: Luer-lock applicator — Applicator for instillation
  Arms: Treatment Group 1: HTX-011; Treatment Group 2: Saline Placebo
Device: Vial access device — Device for withdrawal of drug product
  Arms: Treatment Group 1: HTX-011

SUMMARY:
This is a Phase 3, randomized, double-blind, saline placebo- and active-controlled, multicenter study to evaluate the analgesic efficacy and safety of HTX 011 administered via local administration into the surgical site in subjects undergoing bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo a primary unilateral, distal, first metatarsal bunionectomy with osteotomy and internal fixation under regional anesthesia.
* Has an American Society of Anesthesiologists Physical Status of I, II, or III.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Has had a contralateral foot bunionectomy in the past 3 months.
* Has a planned concurrent surgical procedure (eg, bilateral bunionectomy or collateral procedures on the surgical foot).
* Has other pre existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken any NSAIDs within at least 10 days prior to the scheduled surgery.
* Has taken opioids within 24 hours prior to the scheduled surgery (3 days for long-acting).
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has initiated treatment with medications within 1 month prior to study drug administration that can impact pain control.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* As per subject history and/or medical records, has active infection or is currently undergoing treatment for Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV).
* Has uncontrolled anxiety, psychiatric, or neurological disorder.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse. Note: Subjects with a positive drug screen who are taking an allowed, prescribed medication that is known to result in a positive drug test (eg, amphetamine and dextroamphetamine for attention deficit/hyperactivity disorder, benzodiazepine for anxiety disorder) may be eligible for participation in the study. Subjects taking medical marijuana are not allowed to participate in the study.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half lives.
* Has undergone 3 or more surgeries within 12 months.
* Has a body mass index (BMI) >39 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Springhill Medical Center, Mobile, Alabama
  - Orthopaedic Specialists of North America, PLLC, Mesa, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Trovare Clinical Research, Inc., Bakersfield, California
  - Alliance Research Centers, Laguna Hills, California
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - Optimal Research , LLC, Austin, Texas
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Westside Surgical Hospital, Houston, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Plano Surgical Hospital, Plano, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - EPIC Medical Research, LLC, Murray, Utah
  - Jean Brown Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Yip T, Hu J, Hawn PS, Yamamoto A, Oderda G. HTX-011 effectively reduces postoperative pain intensity and opioid use in the elderly. Pain Manag. 2022 Jan;12(1):45-57. doi: 10.2217/pmt-2021-0043. Epub 2021 Jul 21. PMID 34284613
- [Derived] Viscusi E, Gimbel JS, Pollack RA, Hu J, Lee GC. HTX-011 reduced pain intensity and opioid consumption versus bupivacaine HCl in bunionectomy: phase III results from the randomized EPOCH 1 study. Reg Anesth Pain Med. 2019 May 21:rapm-2019-100531. doi: 10.1136/rapm-2019-100531. Online ahead of print. PMID 31113830

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group 1: HTX-011: HTX 011 (bupivacaine/meloxicam), 60 mg/1.8 mg by instillation.
- Treatment Group 2: Saline Placebo: Saline placebo by instillation.
- Treatment Group 3: Bupivacaine HCI: Bupivacaine HCl without epinephrine, 50 mg by injection.
Period: Overall Study
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Saline Placebo | Treatment Group 3: Bupivacaine HCI
Started | 157 | 100 | 155
Completed | 154 | 99 | 152
Not Completed | 3 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Saline Placebo | Treatment Group 3: Bupivacaine HCI | Total
Number analyzed (Participants) | 157 | 100 | 155 | 412
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 133 | 92 | 139 | 364
  >=65 years | 24 | 8 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (14.47) | 47.3 (12.83) | 45.5 (14.79) | 46.9 (14.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 86 | 132 | 356
  Male | 19 | 14 | 23 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 32 | 49 | 128
  Not Hispanic or Latino | 110 | 68 | 106 | 284
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 8 | 2 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 24 | 12 | 22 | 58
  White | 123 | 86 | 128 | 337
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 157 | 100 | 155 | 412

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores With Activity (NRS-A) Through 72 Hours Postsurgery (AUC0-72), Compared With Saline Placebo.
Description: Pain intensity is assessed using an 11-point NRS (0-10) where 0 represents "no pain" and 10 represents "worst pain imaginable" (using windowed worst observation carried forward to adjust for opioid rescue medication use). The theoretical range of AUC0-72 is 0-720. The prescribed activity for NRS-A is sitting with the plantar surface of the ball of the surgically attended foot touching the floor (no weight bearing).
Time Frame: 72 hours
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Saline Placebo
Number analyzed (Participants) | 157 | 100
pain intensity score*hr | 323.29 (182.641) | 445.34 (155.792)
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 2: Saline Placebo; Test type: Superiority; p < 0.0001, ANOVA; Least Squares Mean Difference (LSMD) = -122.05, 95% CI 2-sided [-163.76 to -80.34], Standard Error of Mean 21.217

2. Secondary Outcome: Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) Pain Intensity Scores With Activity (NRS-A) Through 72 Hours Postsurgery (AUC0-72), Compared With Bupivacaine HCl.
Description: as for outcome 1
Time Frame: 72 hours
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 3: Bupivacaine HCI
Number analyzed (Participants) | 157 | 155
pain intensity score*hr | 323.29 (182.641) | 393.45 (153.756)
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 3: Bupivacaine HCI; Test type: Superiority; p = 0.0002, ANOVA; Least Squares Mean Difference (LSMD) = -70.16, 95% CI 2-sided [-107.07 to -33.25], Standard Error of Mean 18.777

3. Secondary Outcome: Mean Total Postoperative Opioid Consumption (in Morphine Equivalents) for HTX 011 Compared With Saline Placebo.
Time Frame: 72 hours
Population: ITT Population
Measure: Mean (Standard Deviation); unit: IV milligram morphine equivalent (MME)
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Saline Placebo
Number analyzed (Participants) | 157 | 100
IV milligram morphine equivalent (MME) | 18.80 (19.801) | 30.06 (21.016)
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 2: Saline Placebo; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Subjects Who Are Opioid-free for HTX-011 Compared With Bupivacaine HCl.
Time Frame: 72 hours
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 3: Bupivacaine HCI
Number analyzed (Participants) | 157 | 155
Participants | 45 | 17
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 3: Bupivacaine HCI; Test type: Superiority; p = 0.0001, Fisher Exact; Risk Difference (RD) = .177, 95% CI 2-sided [.085 to .265]

5. Secondary Outcome: Mean Total Postoperative Opioid Consumption (in Morphine Equivalents) for HTX 011 Compared With Bupivacaine HCl.
Time Frame: 72 hours
Population: ITT Population
Measure: Mean (Standard Deviation); unit: IV milligram morphine equivalent (MME)
Groups:
- Treatment Group 3: Bupivacaine HCl: Bupivacaine HCl without epinephrine, 50 mg by injection.
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 3: Bupivacaine HCl
Number analyzed (Participants) | 157 | 155
IV milligram morphine equivalent (MME) | 18.80 (19.801) | 25.09 (21.553)
Statistical Analysis 1: Comparison: Treatment Group 1: HTX-011 vs Treatment Group 3: Bupivacaine HCl; Test type: Superiority; p = 0.0022, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 42 days.
Description: For each Preferred Term (PT), subjects are included only once, even if they experienced multiple events in that PT.
Groups:
- Treatment Group 2: Saline Placebo: Saline placebo by instillation.
  1 subject was randomized to bupivacaine HCl, but received saline placebo. (Ie, ITT = 100 and Safety population = 101).
Arm/Group | Treatment Group 1: HTX-011 | Treatment Group 2: Saline Placebo | Treatment Group 3: Bupivacaine HCl
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/101 | 1/154
Serious Adverse Events (participants affected / at risk) | 3/157 | 1/101 | 3/154
Other Adverse Events (participants affected / at risk) | 111/157 | 70/101 | 112/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1: HTX-011 (N=157) | Treatment Group 2: Saline Placebo (N=101) | Treatment Group 3: Bupivacaine HCl (N=154)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis postoperative (Vascular disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1: HTX-011 (N=157) | Treatment Group 2: Saline Placebo (N=101) | Treatment Group 3: Bupivacaine HCl (N=154)
Nausea (Gastrointestinal disorders) | 59 | 44 | 70
Dizziness (Nervous system disorders) | 34 | 18 | 36
Incision site oedema (Injury, poisoning and procedural complications) | 27 | 13 | 22
Vomiting (Gastrointestinal disorders) | 23 | 19 | 33
Headache (Nervous system disorders) | 22 | 10 | 20
Incision site erythema (Injury, poisoning and procedural complications) | 20 | 8 | 18
Post procedural contusion (Injury, poisoning and procedural complications) | 19 | 13 | 18
Bradycardia (Cardiac disorders) | 12 | 6 | 12
Impaired healing (General disorders) | 10 | 1 | 6
Constipation (Gastrointestinal disorders) | 9 | 7 | 18
Muscle twitching (Musculoskeletal and connective tissue disorders) | 9 | 5 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 6 | 1
Sinus arrhythmia (Cardiac disorders) | 6 | 6 | 10
Dysgeusia (Nervous system disorders) | 4 | 6 | 6
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 | 4 | 8
Tinnitus (Ear and labyrinth disorders) | 2 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT03295721/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT03295721/SAP_001.pdf